CLINICAL TRIAL: NCT04089137
Title: Alcohol and Violence Prevention for College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Arizona State University (Other); Medical University of South Carolina (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Amanda Gilmore, Assistant Professor, Mark Chaffin Center for Healthy Development and Department of Health Policy and Behavioral Sciences, School of Public Health, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H20066
Record Dates: First submitted 2019-08-27; First posted 2019-09-13 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Drinking; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will receive an online intervention targeting alcohol misuse and sexual assault among college students. This will include a personalized normative feedback approach. In the first part of the study, there will be an open pilot (1 arm) and in the second part of the study there will be a control condition (2 arms - intervention + control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This is an assessment only control condition.
- Positive Change (+Change) (Experimental): This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse and sexual assault. This intervention targets alcohol use, sexual assault victimization risk, sexual assault perpetration, and bystander intervention and is tailored by gender and sexual orientation.
  Interventions: Behavioral: Positive Change (+Change)

INTERVENTIONS:
Behavioral: Positive Change (+Change) — This is an integrated social norms-based personalized feedback intervention for college students targeting alcohol misuse and sexual assault. This intervention targets alcohol use, sexual assault victimization risk, sexual assault perpetration, and bystander intervention and is tailored by gender and sexual orientation.
  Arms: Positive Change (+Change)

SUMMARY:
Heavy episodic drinking and sexual assault (SA) are problematic on college campuses. This project will adapt already developed interventions targeting alcohol use and SA to a mHealth format and involve content that incorporates federal guidelines and CDC recommendations to integrate both bystander intervention and risk reduction content with new innovative personalized content for each risk group (cis-gender heterosexual men, cis-gender heterosexual women, and sexual/gender minorities). Alpha testing with key stakeholders, an open pilot trial, and a randomized pilot trial will be conducted to establish acceptability and to estimate sample size for a larger randomized controlled trial.

DETAILED DESCRIPTION:
Specific aims are as follows:

Aim 1 (Stage IA): Modify Alcohol and Sexual Assault Prevention (ASAP) content to an eHealth format to include personalized content for each risk group (1. cisgender heterosexual men; 2. cisgender heterosexual women; and 3. sexual and gender minorities).

Aim 1a: Assess normative behaviors (n = 500) regarding alcohol use and SA for feedback.

Aim 1b: Adapt and assess initial acceptability of a workbook version of the intervention content among key stakeholders (college administrators and students from each risk group [n=5 from each group]).

Aim 2 (Stage IB): Open Pilot Trial. Obtain usability of ASAP among 30 students who engage in HED (10 from each risk group) in an open pilot trial.

Aim 3 (Stage IB): A pilot to assess effect size and variability for planning a randomized trial in the future. Randomize students who engage in HED to ASAP or control condition to observe preliminary effect sizes and estimate the variability using a 3-month follow-up. Sample size was determined to estimate the variability within a reasonable margin of error. This calculation also accounted the low base rates of SA and 20% attrition. This led to a sample size of 162 students (n=54 from each risk group).

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* Current student at university of study
* Valid email address at university of study
* Endorse engaging in heavy episodic drinking at least once in the past month on the screening survey

Exclusion Criteria:

* There are no exclusion criteria other than not meeting inclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K Gilmore, PhD, Principal Investigator — Georgia State University
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - Georgia State University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data, only de-identified data.

REFERENCES:
- [Derived] Gilmore AK, Leone RM, Oesterle DW, Davis KC, Orchowski LM, Ramakrishnan V, Kaysen D. Web-Based Alcohol and Sexual Assault Prevention Program With Tailored Content Based on Gender and Sexual Orientation: Preliminary Outcomes and Usability Study of Positive Change (+Change). JMIR Form Res. 2022 Jul 22;6(7):e23823. doi: 10.2196/23823. PMID 35867393

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Positive Change (+Change)
Started | 82 | 83
Completed | 82 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Positive Change (+Change) | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (1.59) | 20.2 (1.66) | 20.35 (1.62)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Cisgender heterosexual woman | 27 | 27 | 54
  Cisgender heterosexual man | 29 | 28 | 57
  Sexual or gender minority | 26 | 28 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 21 | 45
  Not Hispanic or Latino | 58 | 60 | 118
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 1 | 2 | 3
  Asian | 6 | 7 | 13
  Black or African American | 1 | 2 | 3
  White | 63 | 58 | 121
  More than One Race | 5 | 4 | 9
  Other | 5 | 6 | 11
  Prefer not to Answer | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 83 | 165
Enrolled in the study before the COVID-19 pandemic [Count of Participants; unit: Participants] | 38 | 49 | 87

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Enrollment and Recruitment
Description: Feasibility of enrollment recruitment was assessed by the number of anticipated participants enrolled in the study
Time Frame: within 2 year recruitment period
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Positive Change (+Change)
Number analyzed (Participants) | 82 | 83
Participants | 82 | 83

2. Primary Outcome: Feasibility of Retention
Description: Feasibility of retention was assessed by the number of participants retained in the study
Time Frame: within 3 months of baseline participation
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Positive Change (+Change)
Number analyzed (Participants) | 82 | 83
Participants | 71 | 70

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the 3-month data were collection period.
Arm/Group | Control | Positive Change (+Change)
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04089137/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04089137/SAP_002.pdf
  • Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT04089137/ICF_000.pdf